CLINICAL TRIAL: NCT05866536
Title: Repeat BCG Vaccinations for the Treatment of New Onset Type 1 Diabetes in Children Age 8-<18 Years
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Denise Louise Faustman, MD, Director of the Immunobiology Laboratory, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019P002835-RO
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus; Type 1 Diabetes; Diabetes type1; Autoimmune Diabetes
Keywords: Diabetes Mellitus; Type One Diabetes Mellitus; Type I Autoimmune Diabetes Insulin Dependent Diabetes Mellitus 1 IDDM
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bacillus Calmette-Guérin (Experimental): 2 BCG vaccinations spaced 4 weeks apart at the beginning of the trial
  Interventions: Biological: Bacillus Calmette-Guérin
- Saline Injection (Placebo Comparator): 2 placebo injections spaced 4 weeks apart at the beginning of the trial
  Interventions: Biological: Saline Injection

INTERVENTIONS:
Biological: Bacillus Calmette-Guérin — 2 BCG vaccinations spaced 4 weeks apart at the beginning of the trial
  Other Names: BCG
  Arms: Bacillus Calmette-Guérin
Biological: Saline Injection — 2 BCG vaccinations spaced 4 weeks apart at the beginning of the trial
  Arms: Saline Injection

SUMMARY:
The purpose of this study is to investigate if repeat bacillus Calmette-Guérin (BCG) vaccinations can confer a beneficial immune and metabolic effect in new onset pediatric Type 1 diabetes.

DETAILED DESCRIPTION:
Published Phase I data on repeat BCG vaccinations in long term adult type 1 diabetics showed specific death of some of the disease causing bad white blood cells and also showed a short and small pancreas effect of restored insulin secretion. The BCG vaccine also had beneficial metabolic effects that resets the utilization of sugars and significantly improves blood sugars by stably lowering HbA1c values for up to 8 years in subjects in the treatment group and not in the placebo group. In this new onset Phase II Pediatric study, the investigators will attempt to test if even more significant effects can be seen in a new onset pediatric population.

Eligible volunteers will either be vaccinated with BCG twice, one month apart or receive a placebo treatment. Both groups will be followed for five years.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetic subjects diagnosed more than 3 months ago and less than 12 months ago at the time of randomization.
* Male or female, age 8 - <18 years at the time of the screening visit and <18 at the time of randomization.
* HIV antibody negative at the time of the screening visit.
* Human chorionic gonadotropin (hCG) negative at the time of the screening visit, if female.
* M. tuberculosis (TB) negative using a QuantiFERON-TB test prior to randomization, as judged by the Investigator.
* Informed consent and child assent, as age-appropriate, obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial. Legally Acceptable Representative (LAR) of the Subject must sign and date the Informed Consent Form (according to local requirements). The child must sign and date the Child Assent Form or provide oral assent, if required according to local requirements.
* Previously diagnosed with type 1 diabetes mellitus (based on clinical judgement and supported by laboratory analysis as per local guidelines) prior to study enrollment by WHO/ADA diagnostic criteria for glucose levels (FPG = 7.0 mmol/L [126 mg/dL]) or plasma glucose levels 2-hours after 75-gm oral glucose load of = 11.1 mmol/L (200 mg/dL) or a casual plasma glucose >200 mg/dL with symptoms.
* Presence of one or more of the following prior to randomization: antibodies to glutamic acid decarboxylase (GAD), islet cell autoantibody (ICA), protein tyrosine phosphatase-like protein antibodies (IA-2), Insulin autoantibodies (IAA), zinc transporter 8 antibodies (ZnT8).
* Treatment with insulin prior to the screening visit, as judged by the Investigator.
* Ability and willingness to adhere to the protocol, including performing self-measured plasma glucose profiles (Subject and LAR(s) should be evaluated as a unit), as judged by the Investigator.

Exclusion Criteria:

* Clinically significant abnormal screening CBC and chemistries (excluding glucose), as judged by the Investigator.
* Clinically significant screening creatinine elevations above Grade 1, as judged by the Investigator.
* History of chronic infectious disease, such as HIV or untreated or active hepatitis at the time of the screening visit, as judged by the Investigator.
* History of tuberculosis, positive interferon-gamma release assay (IGRA, also known as the QuantiFERON-TB test), including history of a positive test with a high reactivity to mycobacteria of non-tuberculosis variety, prior to randomization (subjects should not be excluded based on history of false positive tests), as judged by the investigator.
* Current treatment with glucocorticoids (other than intermittent nasal or eye steroids, asthma inhaler, or topical steroids), or disease or condition likely to require high dose steroid or immunosuppressive therapy at the time of the screening visit, as judged by the Investigator. This does not include replacement therapies for conditions such as growth hormone deficiencies, Addison's disease, or hypothyroidism.
* Simultaneous participation in any other clinical trial while enrolled in this clinical trial or participation in another clinical trial within 28 days before the screening visit. Note: Clinical trials do not include non-interventional studies.
* Previous participation in the treatment group in biologic or drug intervention trials for Type 1 Diabetes such as anti-CD3.
* Other active chronic conditions, diseases, and/or treatments associated with increased risk of serious side effects and/or morbidities at the time of the screening visit, as judged by the Investigator. This includes conditions that increase the risk of infections, current immunosuppressive therapies for other autoimmune diseases, or patients with a previous history of severe burns.
* Chronic treatment with aspirin > 160 mg/day or chronic, daily NSAIDs at the time of the screening visit, as judged by the Investigator.
* Current treatment with chronic antibiotics that interfere with BCG viability at the time of the screening visit, as judged by the Investigator.
* History of recurrent ketoacidosis with hospitalizations due to non-compliance at the time of the screening visit, as judged by the Investigator.
* History of keloid formation at the time of the screening visit, as judged by the Investigator.
* History or evidence of chronic kidney disease (serum creatinine > 1.5mg/dL), significant protein in the urine, or other significant and/or active diabetes related complication at the time of the screening visit, as judged by the Investigator.
* Screening BMI of <5th percentile or >95th percentile.
* Screening blood pressure >90th percentile for their age and sex.
* Screening temperature >99.8 F.
* Screening heart rate outside of 50-120 bpm.
* History of active proliferative diabetic retinopathy at the time of the screening visit, as judged by the Investigator.
* History of type 2 diabetes or severe obesity at the time of the screening visit, as judged by the Investigator.
* Age of diabetes onset <1.
* Monogenic diabetes at the time of the screening visit.
* Diabetes secondary to cystic fibrosis at the time of the screening visit.
* Diabetes lacking at least 1 diabetes-specific autoantibody prior to randomization.
* History of significant neuropathy, myocardial infarcts, active psychiatric disease that might preclude travel and long-term participation, dementia, foot ulcers, severe diabetes non-compliance, amputations, or kidney disease at the time of the screening visit, as judged by the Investigator.
* History of medical condition(s) that may impact red blood cell turnover such as polycethemia, chronic anemia, vitamin E infusion, transfusion, sickle cell or thalassemia, vitamin C injections, lead poisoning, uremia, or asplenia at the time of the screening visit, as judged by the Investigator.
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using adequate contraceptive methods (adequate contraceptive measures as required by local regulation or practice) at the time of the screening visit, as judged by the Investigator.
* Living with someone who is immunosuppressed and/or at high risk for infectious diseases (for example, HIV+ or taking immunosuppressive medications for any reason) at the time of the screening visit, as judged by the Investigator.
* Current participation in the Phase I or II BCG clinical trial or other immunotherapy diabetes clinical trials at the time of the screening visit, as judged by the Investigator.
* Currently on or planning to take any type 2 diabetes drug or oral blood sugar lowering medication, as judged by the Investigator
* History of the following at the time of the screening visit, as judged by the Investigator: prior BCG vaccination, positive T-spot tuberculosis test indicating active TB, or a T-spot test showing significant Mycobacteria exposure and/or load that would cause a more severe vaccination site inflammation (subjects should not be excluded based on history of false positive tests).
* Not born in the United States.
* Known or suspected hypersensitivity to trial products or related products at the time of the screening visit, as judged by the Investigator.
* Planning to start or change dosage of a medication known to affect glucose metabolism (e.g. thyroid hormones, corticosteroids), as judged by the Investigator, within 14 days prior to the screening visit.
* Any condition, which, in the opinion of the Investigator, might jeopardize the Subject's safety or compliance with the protocol
* Diagnosis of malignant neoplasms within the last five years prior to the screening visit
* Current hypoglycemic unawareness or recurrent severe hypoglycemic episodes at the time of the screening visit, as judged by the Investigator.
* More than one episode of diabetic ketoacidosis requiring hospitalization within the last 90 days prior to the screening.
* Treatment with any medication for the indication of diabetes other than stated in the inclusion criteria in a period of 90 days before screening, as judged by the Investigator.
* History of lupus at the time of the screening visit.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c values | 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, and 5 years after initial BCG/placebo injection
  A change in hemoglobin A1c (HbA1c) values for new onset pediatric type 1 diabetics compared to self.

SECONDARY OUTCOMES:
Change in C-peptide | 1, 2, 3, 4, and 5 years after initial BCG/placebo injection
  A change of fasting or stimulated C-peptide (as an analog for endogenous insulin) in the blood compared to self.
Change in insulin usage | 1, 2, 3, 4, and 5 years after initial BCG/placebo injection
  A change in insulin usage with IDAA1c calculation (adjusting for weight and HbA1c) compared to self.

OTHER OUTCOMES:
Exploratory: Change in hypoglycemia | 1, 2, 3, 4, and 5 years after initial BCG/placebo injection
  A change in hypoglycemic episodes or the magnitude of blood sugar fluctuations compared to self.

CONTACTS AND LOCATIONS:
Overall Officials: Denise L Faustman, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Immunobiology Labs CNY 149, Charlestown, Massachusetts, United States

REFERENCES:
- See also: Faustman Lab Research Website — http://www.faustmanlab.org/